CLINICAL TRIAL: NCT02621658
Title: Clear Liquid vs Liberalized Diet in Preparation for Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: San Antonio Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Luis X. Velez-Colon, MD, Gastroenterology Fellow(PGY5), San Antonio Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Bowel Prep Protocol
Record Dates: First submitted 2015-11-23; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Colonoscopy; Adenoma Detection Rate; Bowel Preparation; Time to Cecal Intubation
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clear Liquid Diet (Active Comparator): Clear Liquid Diet the day before colonoscopy.
  Interventions: Other: Clear Liquid Diet
- Full Liquid Diet (Experimental): Full Liquid Diet the day before colonoscopy.
  Interventions: Other: Full Liquid Diet

INTERVENTIONS:
Other: Clear Liquid Diet — Patients will be allowed to consume clear soft drinks like ginger ales, Sprite®, 7-Up®, Gatorade®, Kool Aid®. They can also have strained fruit juices like apple, white grape juice and lemonade, and water, tea and coffee without milk or non-dairy creamer. Patient in this arm will also be allowed to have low-sodium chicken or beef broth , in addition to non-red hard candies, Jell-O®, and popsicles.
  Arms: Clear Liquid Diet
Other: Full Liquid Diet — Patients will be allowed to consume a Full Liquid Diet, including nutritional supplements(Ensure®, Boost®, Glucerna®), strained cereals(like cream of wheat or strained oatmeal) and vegetables, purred fruit without seeds or pulp, milk, plain ice cream or yogurt, sherbet, coffee with cream, and tea.
  Arms: Full Liquid Diet

SUMMARY:
Colorectal cancer is the third most common cancer diagnosed in both men and women in the United States. The death rate from this disease, however, has been decreasing over the last 20 years. Early detection and removal of pre-malignant polyps is considered to be at the core of this change. At the same time, polyp detection is highly dependent on an adequate bowel preparation. Froehlich, et al., found that poor bowel preparation is associated with longer colonoscopy times, more difficult procedures and a higher rate of incomplete procedures(2).

Although a Clear Liquid Diet is usually the prescribed diet in most bowel preparation regimes, several studies have shown similar results with less restrictive diets.

Based on the hypothesis that a Full Liquid Diet(FLD) is not inferior to a Clear Liquid Diet(CLD), investigators plan to conduct a prospective, randomized trial, in order to compare these dietary interventions. The investigators and endoscopists will be blinded to patient's diet group.

Researchers aim to investigate if diet liberalization to a Full Liquid Diet(FLD) is associated with similar bowel cleansing as compared with a Clear Liquid Diet(CLD). Investigators will compare the performance of these dietary interventions regarding adenoma detection rates(ADR), time to cecal intubation(TCI), and colonoscope withdrawal time. In addition, the investigators want to assess whether patient's Compliance and Satisfaction is similar or superior in the experimental group vs the control group.

DETAILED DESCRIPTION:
The purpose of this study is to investigate if a Full Liquid Diet is not inferior to a Clear Liquid Diet in preparation for Screening Colonoscopy. Based on the data presented above, the investigators hypothesize that a Full Liquid Diet will be better tolerated by participants and will not adversely affect colonoscopy outcomes in terms of bowel cleansing(BC), adenoma detection rate(ADR), time to cecal intubation(TCI).

The results of this study may help guide dietary interventions in preparation for Colonoscopy in the Department of Defense(DOD) Military Treatment Facilities.

The relationship between adequate colon cleansing and adenoma detection rate(ADR) has been already established. Almost 25% of patients, however, have a poor bowel preparation at the time of Colonoscopy(1). After reviewing 5832 colonoscopies, Froehlich, et al., found that poor bowel preparation is associated with longer colonoscopy times, more difficult procedures and a higher rate of incomplete procedures(2).

Among other causes, bowel cleansing is affected by purgative selection and timing of administration, compliance with recommended pre-procedural diet and compliance with purgative administration. Recently, it has been found that the classically recommended clear liquid diet(CLD) is not indispensable for adequate bowel prep. Stolpman, et. al, found that a low-residue diet is non-inferior to clear liquid diet(CLD), in a group of 201 patients(3). Similarly, Melicharkova, et al, found that the bowel cleansing efficacy of a low-residue breakfast, the day before colonoscopy, was comparable with a clear liquid diet(CLD) in a sample of 213 patients administered a low volume purgative in preparation for colonoscopy(4). They also found a statistically significant difference in the level of patient's acceptance of the low-residue diet.

A group from South Korea, led by Dr. Jung Yoon, found similar rates of bowel cleansing in patient undergoing afternoon colonoscopy, when offered Regular Diet(5). A study, in a small study population, presented as an abstract at the American College of Gastroenterology Conference in 2011, reported comparable bowel cleansing, polyp detection rate, and colonoscopy times in patients allowed a full liquid diet before the procedure(6). Taken together, these studies show that a clear liquid diet may not be necessary in order to obtain a good bowel cleanse in preparation for colonoscopies performed in the outpatient setting.

A clear liquid diet is still the recommended diet, however, before this procedure.

Given the diverse population served at Military Treatments Facilities across the United States, and abroad, the investigators aim to investigate if diet liberalization to a Full Liquid Diet(FLD) is associated with similar bowel cleansing as compared with a Clear Liquid Diet(CLD). In addition, the investigators will compare the performance of these diets regarding adenoma detection rates(ADR), time to cecal intubation(TCI), withdrawal time, and patient satisfaction.

This study will be conducted as a prospective, randomized trial. The investigators and endoscopists will be blinded to patient's diet group.

Patients 50 y/o, or older, undergoing screening colonoscopy will be offered participation in the study.

If written, informed consent is obtained, participants will be randomized to (A)Control Group or (B) Study Group(in a 1:1 fashion). Study randomization will be performed by using serially numbered envelopes containing instructions for CLD or FLD. The control group will be allowed to have a Clear Liquid Diet the day before colonoscopy and the Study Group will be allowed to have a Full Liquid Diet the day before colonoscopy. These envelopes will be prepared in duplicates. One envelope will be provided to the participant and one envelope will be maintained, sealed, by the study group.

Study participants will complete a Bowel Preparation consisting of bisacodyl 10mg per mouth x1(at noon, the day before colonoscopy) and 4L Polyethylene Glycol solution(split dose). Subjects will drink 2 L of Polyethylene Glycol at 17:00 the day before colonoscopy and the other 2 L at 04:00, the morning prior to colonoscopy.

They will follow one of the diets described above, based on randomization, and will present to the BAMC Gastroenterology Clinic for Colonoscopy. Before the procedure, subjects will be administered a questionnaire in order to assess their compliance, tolerability and satisfaction with the diet. Research team and Endoscopists will also be blinded to these questionnaires until the data collection process has finished.

Colonoscopy will be performed in the usual fashion. Endoscopists will assess the level of subject's colon cleansing by means of the Boston Bowel Preparation Scale(7). Time to Cecal Intubation and Colonoscope Withdrawal Time will be documented, as is currently done at the BAMC Gastroenterology Clinic.

Adenoma Detection Rates(number of screened patients with at least one adenoma divided by total number of patients screened with colonoscopy) will be calculated.

Investigators will compare Bowel Prep Quality/Colon Cleansing, Time to Cecal Intubation, ADR, and Patient's Compliance and Satisfaction with the bowel preparation between the two groups.

Primarily, the investigators want to assess whether Bowel Prep Quality/Colon Cleansing and ADR for the experimental group is non-inferior to Bowel Prep Quality and ADR for the control group. In addition, the investigators will asses whether participant's Compliance and Satisfaction is similar or superior in the experimental group vs the control group.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic patients 50 years old or older, undergoing screening colonoscopy and willing to participate in the study will be included, after obtaining informed/written consent.

Exclusion Criteria:

* Symptomatic patients, patients with indications for therapeutic colonoscopy, like for example, rectal bleeding or with a prior diagnosis requiring evaluation with colonoscopy(Prior diagnosis of colon polyps, Iron-deficiency Anemia, Inflammatory Bowel Disease, Colorectal Cancer, Chronic diarrhea, Abnormal Imaging) will be excluded from participation. Please note that patients with Iron-deficiency Anemia will not be excluded from the study, based solely on this diagnosis, if they have an indication, otherwise, for Screening Colonoscopy.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Bowel Preparation | At the time of Colonoscopy
  This will be assessed using the Boston Bowel Preparation Scale
Time to Cecal Intubation | During Colonoscopy
Colonoscope Withdrawal time | During Colonoscopy
  Time elapsed since the endoscopist starts withdrawing the colonoscope, after reaching the cecum, until the completion of the test.
Adenoma Detection Rate | During Colonoscopy
  Number of patients with at least one adenoma, divided by total number of patients aged 50 years or older screened with colonoscopy

SECONDARY OUTCOMES:
Patient compliance | Before Colonoscopy
  Will be measured using a questionnaire
Patient satisfaction | Before Colonoscopy
  Will be measured using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Luis X Velez-Colon, MD, Principal Investigator — San Antonio Military Medical Center

REFERENCES:
- [Background] Harewood GC, Sharma VK, de Garmo P. Impact of colonoscopy preparation quality on detection of suspected colonic neoplasia. Gastrointest Endosc. 2003 Jul;58(1):76-9. doi: 10.1067/mge.2003.294. PMID 12838225
- [Background] Stolpman DR, Solem CA, Eastlick D, Adlis S, Shaw MJ. A randomized controlled trial comparing a low-residue diet versus clear liquids for colonoscopy preparation: impact on tolerance, procedure time, and adenoma detection rate. J Clin Gastroenterol. 2014 Nov-Dec;48(10):851-5. doi: 10.1097/MCG.0000000000000167. PMID 25296243
- [Background] Jung YS, Seok HS, Park DI, Song CS, Kim SE, Lee SH, Eun CS, Han DS, Kim YS, Lee CK. A clear liquid diet is not mandatory for polyethylene glycol-based bowel preparation for afternoon colonoscopy in healthy outpatients. Gut Liver. 2013 Nov;7(6):681-7. doi: 10.5009/gnl.2013.7.6.681. Epub 2013 Aug 14. PMID 24312709
- [Background] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Background] Melicharkova A, Flemming J, Vanner S, Hookey L. A low-residue breakfast improves patient tolerance without impacting quality of low-volume colon cleansing prior to colonoscopy: a randomized trial. Am J Gastroenterol. 2013 Oct;108(10):1551-5. doi: 10.1038/ajg.2013.21. PMID 24091500
- [Background] Full Liquid Diet vs Clear Liquid Diet for Colonoscopy Preparation: Preliminary Results. Gutkin E, et. al. ACG2011; Abstract P412
- [Background] Calderwood AH, Jacobson BC. Comprehensive validation of the Boston Bowel Preparation Scale. Gastrointest Endosc. 2010 Oct;72(4):686-92. doi: 10.1016/j.gie.2010.06.068. PMID 20883845
- [Background] Agresti A, Coull BA, Approximate is better than "exact" for interval estimation of binomial proportions, The American Statistician 52:119-126, 1998.
- [Background] Jones B, Jarvis P, Lewis JA, Ebbutt AF. Trials to assess equivalence: the importance of rigorous methods. BMJ. 1996 Jul 6;313(7048):36-9. doi: 10.1136/bmj.313.7048.36. PMID 8664772